CLINICAL TRIAL: NCT02550912
Title: A Pilot Study Evaluating the Effect of Vitamin D on Clinical Outcome in Autistic Children
Brief Title: A Study Evaluating the Effect of Vitamin D on Clinical Outcome in Autistic Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sarah Farid Mohamed Fahmy, Assistant lecturer in clinical pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PhD(NO.18)
Record Dates: First submitted 2015-09-12; First posted 2015-09-16 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Cholecalciferol; High Fructose Corn Syrup

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D group (Active Comparator): Patients will receive vitamin D drug with generic name: V drops manufactured by Medical Union Pharmaceuticals, Egypt Dosage form: liquid drops Dosage, frequency, and Duration:1000 international units per day for 3 months then 1000 international units per 25 pounds per day for another 3 months.
  Interventions: Drug: Vitamin D3
- Placebo group (Placebo Comparator): Patients will receive glucose syrup same taste and color as vitamin D3 drops with same dosage regimen to vitamin D group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — vitamin D drops for paediatrics
  Other Names: vitamin D drops
  Arms: Vitamin D group
Other: Placebo — glucose syrup with same taste and color to vitamin D3 drops
  Other Names: glucose syrup
  Arms: Placebo group

SUMMARY:
The purpose of this study to determine whether high dose vitamin D has positive effect on behavior of autistic children.

DETAILED DESCRIPTION:
Double blinded placebo controlled study to determine effect of two different doses of vitamin D on Behavioral domains in autistic children.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfill fourth edition of Diagnostic and statistical manual of mental Disorders (DSM 4th) criteria for autism

Exclusion Criteria:

* Patients who had seizures within the past year or History of kidney or liver disease or Taking the following medications or supplements that may affect vitamin D level (as antiepileptic, corticosteroids or immunosuppressant) were excluded from the study. None of the study participants received vitamin D or calcium therapy in the past 6 months and there were no change in children's treatment regimen (including medications) within 1 month prior to the study.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Effect of vitamin D on changes in behavioral measures (Childhood autism rating scale) | At baseline, 12 weeks ,24 weeks
Effect of vitamin D on changes in behavioral measures (autism treatment evaluation checklist) | At baseline, 12 weeks ,24 weeks

SECONDARY OUTCOMES:
Effect of vitamin D on calcium level | At baseline, 12 weeks ,24 weeks
Effect of vitamin D on phosphorous level | At baseline, 12 weeks ,24 weeks
Effect of vitamin D on alkaline phosphatase level | At baseline,12 weeks ,24 weeks
Effect of vitamin D on parathyroid hormone level | At baseline,12 weeks ,24 weeks
Effect of vitamin D on liver function test (alanine transaminase and aspartate transaminase) | At baseline, 12 weeks ,24 weeks
Effect of vitamin D on kidney function test (Blood urea nitrogen and serum creatinine) | At baseline, 12 weeks ,24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: sarah f mohamed fahmy, masters, Principal Investigator — assistant lecturer clinical pharmacy ainshams university; nagwa A sabri, professor, Study Director — professor in clinical pharmacy Ainshams university; manal H elhamamsy, professor, Study Director — professor in clinical pharmacy Ainshams university; mohamed A elsawi, professor, Study Director — professor in pediatrics and genetics ainshams university; osama k zaki, consultant, Study Director — medical consultant in paediatrics and genetics unit ainshams university
Locations (1):
- Faculty of Pharmacy AinShams University, Cairo, Egypt